CLINICAL TRIAL: NCT06421935
Title: An Open Label, Multicenter, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of the PARP1 Inhibitor M9466 Alone or in Combination in Participants With Advanced Solid Tumors
Brief Title: M9466 Alone or in Combination in Advanced Solid Tumors (DDriver 501)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS202659_0001; 2024-513492-41-00 (Other: EU CTR)
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: PARP inhibitor; castration-resistant Prostate cancer; ovarian cancer; Abiraterone Acetate
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Abiraterone Acetate; abiraterone; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- M9466 plus Tuvusertib (Experimental)
  Interventions: Drug: M9466; Drug: Tuvusertib
- M9466 Monotherapy (Experimental)
  Interventions: Drug: M9466
- M9466 with AA-P(abiraterone acetate and prednisone or prednisolone) (Experimental)
  Interventions: Drug: M9466; Drug: Abiraterone acetate; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: M9466 — Participants will be administered M9466 orally.
  Other Names: HRS-1167;
Drug: Tuvusertib — Participants will be administered Tuvusertib orally.
  Other Names: Substance code MSC2584415A; also known as M1774, VXc-400, or VR 1363004
  Arms: M9466 plus Tuvusertib
Drug: Abiraterone acetate — Participants will be administered with Abiraterone acetate orally.
  Other Names: Abiraterone
  Arms: M9466 with AA-P(abiraterone acetate and prednisone or prednisolone)
Drug: Prednisone/Prednisolone — Participants will be administered with prednisone/prednisolone orally.
  Arms: M9466 with AA-P(abiraterone acetate and prednisone or prednisolone)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamic profile of M9466 with and without tuvusertib or an ARPi and early signs of clinical activity of M9466 with tuvusertib in participants with advanced solid tumors. Study details include: Study/Treatment Duration: Participants will be treated until disease progression, death, discontinuation, or End of Study. Visit Frequency: Every week in the first 2 cycles, followed by every 3 weeks in the subsequent cycles. An End of Treatment Visit and Safety Follow-up/Discontinuation Visit are scheduled after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Module 1 Part A and Module 2 Part A1: Locally advanced or metastatic disease that is refractory to standard therapy or for which no standard therapy is judged appropriate by the Investigator
* Module 1 Part A2: Histologically or pathologically confirmed advanced or metastatic CRPC or EOC
* Eastern Cooperative Oncology Group Performance Status less than or equal to (<=) 1
* Life expectancy of more than 6 months
* Have adequate hematologic function
* Participants who received chemotherapy, extensive radiotherapy, biological therapy (e.g. antibodies) or investigational agents will have a washout period of 4 weeks (6 weeks for nitrosourea, mitomycin-C) or 5 half-lives whichever is shorter, prior to starting study intervention with M9466 (± tuvusertib)
* Module 3 Part A1:

  * Histologically or pathologically confirmed diagnosis of prostate cancer
  * Metastatic disease documented by positive bone scan or metastatic lesions on CT or MRI
  * Participants with Metastatic Castration-Resistant Prostate Cancer (mCRPC) or metastatic hormone-sensitive prostate cancer (mHSPC) are allowed. For mCRPC, serum testosterone levels ≤ 50 /dL (≤ 1.75 nmol/L).
  * Ongoing ADT with a GnRH agonist or antagonist for participants who have not undergone bilateral orchiectomy must be initiated before first dose and must continue throughout the study.
  * Candidate for treatment with ·abiraterone acetate.
  * Prior anticancer therapy allowed for mHSPC or mCRPC
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Persistence of Adverse Events related to any prior treatments that have not recovered to Grade less than 1 by NCI Common Terminology Criteria for Adverse Events- v5.0 unless AEs are clinically nonsignificant and/or stable on supportive therapy in the opinion of the Investigator (e.g. neuropathy or alopecia)
* Participant has a history of additional malignancy within 5 years before the date of enrollment other than disease under study (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertropia, or malignancy that in the opinion of the Investigator, with concurrence of the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years)
* Participants with known brain metastases, except if clinically controlled, which is defined as individuals with Central Nervous System (CNS) tumors that have been treated, are asymptomatic and who have discontinued steroids (for the treatment of CNS tumors) for more than 28 days
* Serious Gastrointestinal bleeding within 3 months, refractory nausea and vomiting, uncontrolled diarrhea, known malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes, other chronic gastrointestinal disease (including exocrine pancreatic insufficiency requiring pancreatic enzyme replacement therapy), and/or other situations that may preclude adequate absorption of oral medications
* Cerebrovascular accident or stroke
* Module 3 only:

  * Current evidence of any of the following:

    1. Any medical condition that would make prednisone (or equivalent) use contraindicated.
    2. Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone (or equivalent) once daily.
  * History of uncontrolled pituitary or adrenal dysfunction
  * Hypokalemia
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Module 1 Part A1 and Part A2: Number of Participants With Treatment-Emergent Adverse Events (TEAE), and Treatment-related AEs (TRAEs) | Time from first treatment up to 30 days after end of study intervention (approximately assessed up to 20 months)
Module 1 Part A1 and Part A2: Number of Participants with Dose Limiting Toxicity (DLT)-like events | Day 1 up to Day 21 of Cycle 1 (each cycle is of 21 days)
Module 2 Part A1: Pharmacokinetic (PK) Plasma Concentrations of M9466 | Cycle 1 Day 1 (C1D1), C1D8 and C1D15
Module 2 Part A2: Number of Participants With Treatment-Emergent Adverse Events (TEAE), and Treatment-related AEs (TRAEs) | Time from first treatment up to 30 days after end of study intervention (approximately assessed up to 20 months)
Module 3 Part A1: Number of Participants With Treatment-Emergent Adverse Events (TEAE), and Treatment-related AEs | Time from first treatment up to 30 days after end of study intervention
Module 3 Part A1: Number of Participants with Dose Limiting Toxicity (DLT)-like Events | Day 1 up to Day 21 of Cycle 1(each cycle is of 21 days)

SECONDARY OUTCOMES:
Module 1 Part A1 and Part A2, Module 2 Part A1 and A2 and Module 3 Part A1: Pharmacokinetic (PK) Plasma Concentrations of M9466 and Tuvusertib | Module 1 Part A1: C1D1 and C1D5 or C1D6; Module 1 Part A2: C1D1, C1D2, C1D3 or C1D4 and C1D8; Module 2 Part A1: C1D1, C1D8 and C1D15; Module 2 Part A2: C1D1, C1D2 and C1D8, C1D22 and C2D1; Module 2 Part A1: C1D1 and C1D8
Module 1 Part A1 and Part A2, Module 2 Part A2: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (or PCWG3 for prostate cancer) as Assessed by Investigator | Time from first treatment to planned assessment at 12 months
Module 1 Part A1 and Part A2; Module 2 Part A1 : Effect of M9466 in combination with tuvusertib on QTc interval as determined by Digital ECGs | Time from first treatment to planned assessment at 12 months
Module 2 Part A1: Number of Participants With Treatment-Emergent Adverse Events (TEAE), and Treatment-Related AEs | Time from first treatment up to 30 days after end of study intervention (approximately assessed up to 20 months)
Module 2 Part A1 and Part A2: Relative Changes in Pharmacodynamics Markers in Paired Tumor Biopsies | Day 1, Day 8 and Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (20):
- United States (2):
  - NEXT Oncology - PARENT, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Cancer Research SA, Adelaide
  - GenesisCare North Shore (Oncology), St Leonards
- Japan (4):
  - Harasanshin Hospital, Fukuoka
  - National Cancer Center Hospital East - Dept of Experimental Therapeutics, Kashiwa-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - NHO Kumamoto Medical Center - Dept of Urology, Kumamoto
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System - Division of Infectious Diseases, Seoul
- Spain (7):
  - Hospital HM Nou Delfos - START Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, Barcelona
  - Centro Integral Oncologico Clara Campal - Unidad de Fase I-Oncologica, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz - START Madrid FJD - Oncology Phase I, Madrid
  - NEXT Madrid - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html